CLINICAL TRIAL: NCT05654662
Title: A Randomized, Controlled, Examiner-Blind Clinical Study Investigating the Effects of a Dentifrice Containing 67% Sodium Bicarbonate When Used Twice Daily for 12 Weeks on Gingivitis Treatment and Plaque Removal
Brief Title: A Clinical Study Investigating the Effects of a Dentifrice Containing 67% Sodium Bicarbonate When Used Twice Daily for 12 Weeks on Gingivitis Treatment and Plaque Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 300029
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-11

CONDITIONS: Gingivitis; Dental Plaque
MeSH Terms: conditions — Gingivitis; Dental Plaque

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corsodyl Original Dentifrice (Experimental): Participants will be instructed to brush their teeth using test product for at least a minute twice a day (morning and evening) for 12 weeks. Participants will dose the toothbrush provided with a ribbon of paste to cover the brush head (a full brush head) on each brushing occasion.
  Interventions: Drug: Corsodyl Original Dentifrice
- Colgate Cavity Protection Dentifrice (Active Comparator): Participants will be instructed to brush their teeth using reference product for at least a minute twice a day (morning and evening) for 12 weeks. Participants will dose the toothbrush provided with a ribbon of paste to cover the brush head (a full brush head) on each brushing occasion.
  Interventions: Drug: Colgate Cavity Protection Dentifrice

INTERVENTIONS:
Drug: Corsodyl Original Dentifrice — It contains 67% weight/weight (w/w) Sodium Bicarbonate and 0.310% w/w Sodium Fluoride (1400 parts per million [ppm] Fluoride ion [F])
  Arms: Corsodyl Original Dentifrice
Drug: Colgate Cavity Protection Dentifrice — It contains 0.76% w/w Sodium Monofluorophosphate (1000 ppm F) and 0.1% w/w Sodium Fluoride (450 ppm F)
  Arms: Colgate Cavity Protection Dentifrice

SUMMARY:
The main goal of this study is to evaluate and compare the efficacy of an on-market dentifrice containing 67 percent (%) sodium bicarbonate and 0.31% sodium fluoride to a reference regular fluoride dentifrice on treating gingival bleeding and gingival inflammation as well as reducing plaque accumulation in population with gingivitis after 12 weeks use.

DETAILED DESCRIPTION:
This will be a single center, controlled, single blind (examiner blind), randomized, two treatment arm, parallel study in volunteers with clinically measurable levels of gingivitis (defined as those with 10-30% bleeding sites on probing). Approximately 200 participants (100 per group) will be randomized to ensure 188 evaluable participants (94 per group) complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the Participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participant who is willing and able to comply with scheduled visits, treatment plan, and other study procedures.
* A Participant in good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant/relevant abnormalities in medical history or upon oral examination, or condition, that would impact the Participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
* Participant oral health that meets all the following:

At Screening (Visit 1):

1. Participant with at least 20 natural, permanent teeth.
2. Participant with at least 40 evaluable surfaces for MGI, BI, and TPI (An evaluable surface is defined as having 2/3rds of the natural tooth surface gradable for the selected clinical indices. The following should not be included in the evaluable surface count- third molars; fully crowned/extensively restored, grossly carious, orthodontically banded/bonded or abutment teeth; surfaces with calculus deposits which, in the opinion of the clinical examiner, would interfere with the baseline assessments of the selected clinical indices).
3. A participant with plaque-induced gingivitis, in the opinion of the clinical examiner, as confirmed by a gross visual examination at the Screening Visit.

At Baseline (Visit 2):

1. A participant with ongoing hard tissue eligibility and, in the opinion of the clinical examiner, at least 40 evaluable surfaces.
2. A participant with 10% less than (<) bleeding on probing (BOP) < 30%.
3. A participant with mean whole mouth TPI score more than or equal to (>=)1.5.

Exclusion Criteria:

* A participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a sponsor's employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
* A participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* A participant who has any other clinical serious or unstable conditions (such as, cardiovascular diseases, diabetes, liver disorders, and kidney disorders) which could have affected study out comes and/or participant safety.
* A participant who is a pregnant female (self-reported) or is intending to become pregnant over the duration of the study.
* A participant who is a breastfeeding female.
* A participant who is known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* A participant who is unwilling or unable to comply with the lifestyle considerations.
* Participant who is a current smoker or an ex-smoker who stopped within 6 months of Screening.
* Participant who is using smokeless forms of tobacco (such as, chewing tobacco, gutkha, pan containing tobacco, nicotine-based e-cigarettes).
* A participant who is diagnosed xerostomia or is taking any medication that in the view of the investigator is causing xerostomia.
* A participant who has a medical condition which could have directly influenced gingival bleeding.
* A participant who has a bleeding disorder that could have affected study outcomes and/or participant safety.
* A participant who has a recent history (within the last year) of alcohol or other substance abuse.
* A participant who has a severe oral condition (such as, acute necrotizing ulcerative gingivitis or oral or peri-oral ulceration including herpetic lesions) that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant/examiner if they participate in the study.
* Presence of a tongue or lip piercing, or any other oral feature that could interfere with the usage of a toothbrush.

Medication Exclusions At Screening (Visit 1):

1. A participant using any antibiotic medication within 14 days prior to screening or at any time during the study.
2. A participant currently taking an anti-inflammatory medication which, in the opinion of the Investigator, could affect gingival condition.
3. A participant currently taking a systemic medication (such as, anti-inflammatory, anticoagulant, immunosuppressants) or traditional/ herbal remedy which, in the opinion of the Investigator, could affect plaque/ gingival condition (such as, ibuprofen, aspirin, warfarin, cyclosporin, phenytoin, calcium channel blockers).

Medication Exclusions at Baseline (visit 2):

1. A participant who has taken (in the previous 14 days), any antibiotics.
2. A participant who has taken (in the previous 14 days) a systemic medication (such as, anti-inflammatory, anti-coagulant, immunosuppressants) or traditional/ herbal remedy which, in the opinion of the Investigator, could affect plaque/ gingival condition (such as, ibuprofen, aspirin, warfarin, cyclosporin, phenytoin, calcium channel blockers).
3. A participant who has used an antibacterial dentifrice or mouthwash (such as, chlorhexidine) or any oral care product that in the view of the investigator could interfere with plaque formation or measures of gingivitis, in the period between Screening and the Baseline visit.

Periodontal Exclusions

1. A participant who shows signs of periodontitis (one or more sites with probing pocket depths more than [>] 3 mm).
2. A participant who is receiving or has received treatment for periodontal disease (including surgery) within 12 months of Screening.
3. A participant who has gingivitis, which in the opinion of the investigator, is not expected to respond to treatment with an over the counter (OTC) dentifrice.

Dental Exclusions

1. A participant who has active caries that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant if they participate in the study.
2. A participant who has dentures (partial or full).
3. A participant who has an orthodontic appliance (bands, appliances, or fixed/ removable retainers).
4. A participant who received orthodontic therapy within 3 months of Screening.
5. A participant who has numerous restorations in a poor state of repair.
6. A participant who has any dental condition (such as, overcrowding) that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant if they participate in the study.
7. A participant who has had dental prophylaxis within 12 weeks of Screening.
8. A participant who has had teeth bleaching within 12 weeks of Screening.
9. A participant who has high levels of extrinsic stain or calculus deposits, in the opinion of the investigator, that could have interfered with plaque assessments.
10. A participant who has previously been enrolled in this study.
11. A participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bristol, Bristol Dental School and Hospital, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in the United Kingdom.
Pre-assignment Details: A total of 204 participants were screened of which 197 participants were enrolled, and 190 participants were randomized to receive treatment in 2 groups: Test Product group (94 participants) and Reference Product group (96 participants). 14 participants were not randomized (9 participants did not meet study criteria; 2 participants were lost to follow-up; and 3 participants withdrew their consent). A total of 188 randomized participants completed the study.
Groups:
- Test Product (Corsodyl Original Toothpaste): Participants were instructed to dose the toothbrush provided with full ribbon of test product (Corsodyl Original Toothpaste) containing 67 percent (%) weight/weight (w/w) Sodium Bicarbonate and 0.310% w/w Sodium Fluoride and brush their teeth for at least a minute, twice daily (morning and evening) for 12 weeks.
- Reference Product (Colgate Cavity Protection Toothpaste): Participants were instructed to dose the toothbrush provided with full ribbon of reference product (Colgate Cavity Protection Toothpaste) containing 0.76% w/w Sodium Monofluorophosphate and 0.1% w/w Sodium Fluoride and brush their teeth for at least a minute, twice daily (morning and evening) for 12 weeks.
Period: Overall Study
Arm/Group | Test Product (Corsodyl Original Toothpaste) | Reference Product (Colgate Cavity Protection Toothpaste)
Started | 94 | 96
Completed | 92 | 96
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — A death in the family | 1 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat (mITT) Population included all randomized participants who completed at least 1 dose of the study product and had at least 1 post-Baseline clinical performance assessment.
Groups:
- Test Product (Corsodyl Original Toothpaste): Participants were instructed to dose the toothbrush provided with full ribbon of test product (Corsodyl Original Toothpaste) containing 67% w/w Sodium Bicarbonate and 0.310% w/w Sodium Fluoride and brush their teeth for at least a minute, twice daily (morning and evening) for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Test Product (Corsodyl Original Toothpaste) | Reference Product (Colgate Cavity Protection Toothpaste) | Total
Number analyzed (Participants) | 94 | 96 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (12.08) | 39.8 (13.20) | 39.5 (12.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 67 | 136
  Male | 25 | 29 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 94 | 96 | 190
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 4 | 8 | 12
  Asian - Central/South Asian Heritage | 5 | 10 | 15
  Asian - East Asian Heritage | 1 | 2 | 3
  Asian - South East Asian Heritage | 1 | 0 | 1
  White - White/Caucasian/European Heritage | 73 | 71 | 144
  Multiple | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Number of Bleeding Sites at Week 12
Description: The number of bleeding sites was calculated using the bleeding index (BI) assessment. The BI was assessed for all evaluable surfaces (having two-thirds of the natural tooth surface gradable for the assessment) of the facial and lingual/palatal gingiva, 6 sites per tooth (mesiobuccal, buccal, and distobuccal; mesiolingual/palatal, lingual/palatal, and distolingual/palatal). Evaluable tooth sites were probed, and gingival bleeding was assessed for approximately 30 seconds after probing. The number of bleeding sites for each participant was calculated as the number of evaluable tooth sites with bleeding observed immediately on probing or within 30 seconds of probing. Change from Baseline was calculated by subtracting the Baseline value from the value at Week 12. Baseline was defined as Day 0. A negative change from Baseline indicated improvement in gingival bleeding.
Time Frame: Baseline and Week 12
Population: mITT Population. Here, overall number analyzed is defined as the number of participants with data available for analysis of this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: bleeding sites
Arm/Group | Test Product (Corsodyl Original Toothpaste)
Number analyzed (Participants) | 92
bleeding sites | -4.3 (1.44)
Statistical Analysis 1: Comparison: Test Product (Corsodyl Original Toothpaste); Change from Baseline at Week 12 (Test for non-zero within group change from Baseline); Test type: Superiority; p = 0.0032, MMRM

2. Secondary Outcome: Adjusted Mean Change From Baseline in Number of Bleeding Sites at Week 12 (Test Product Versus [vs.] Reference Product)
Description: The number of bleeding sites was calculated using the BI assessment. The BI was assessed for all evaluable surfaces (having two-thirds of the natural tooth surface gradable for the assessment) of the facial and lingual/palatal gingiva, 6 sites per tooth (mesiobuccal, buccal, and distobuccal; mesiolingual/palatal, lingual/palatal, and distolingual/palatal). Evaluable tooth sites were probed, and gingival bleeding was assessed for approximately 30 seconds after probing. The number of bleeding sites for each participant was calculated as the number of evaluable tooth sites with bleeding observed immediately on probing or within 30 seconds of probing. Change from Baseline was calculated by subtracting the Baseline value from the value at Week 12. Baseline was defined as Day 0. A negative change from Baseline indicated improvement in gingival bleeding.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: bleeding sites
Arm/Group | Test Product (Corsodyl Original Toothpaste) | Reference Product (Colgate Cavity Protection Toothpaste)
Number analyzed (Participants) | 92 | 96
bleeding sites | -4.3 (1.44) | 2.3 (1.42)
Statistical Analysis 1: Comparison: Test Product (Corsodyl Original Toothpaste) vs Reference Product (Colgate Cavity Protection Toothpaste); Test type: Superiority; p = 0.0013, Mixed Model with Repeated Measure (MMRM); Adjusted Mean Difference = -6.6, 95% CI 2-sided [-10.6 to -2.6], Standard Error of Mean 2.03 — Adjusted mean difference was calculated as test product minus reference product

3. Secondary Outcome: Adjusted Mean Change From Baseline in Number of Bleeding Sites at Week 3 and Week 6
Description: The number of bleeding sites was calculated using the BI assessment. The BI was assessed for all evaluable surfaces (having two-thirds of the natural tooth surface gradable for the assessment) of the facial and lingual/palatal gingiva, 6 sites per tooth (mesiobuccal, buccal, and distobuccal; mesiolingual/palatal, lingual/palatal, and distolingual/palatal). Evaluable tooth sites were probed, and gingival bleeding was assessed for approximately 30 seconds after probing. The number of bleeding sites for each participant was calculated as the number of evaluable tooth sites with bleeding observed immediately on probing or within 30 seconds of probing. Change from Baseline was calculated by subtracting the Baseline value from the value at each indicated timepoint. Baseline was defined as Day 0. A negative change from Baseline indicated improvement in gingival bleeding.
Time Frame: Baseline, Week 3, and Week 6
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Least Squares Mean (Standard Error); unit: bleeding sites
Arm/Group | Test Product (Corsodyl Original Toothpaste)
Number analyzed (Participants) | 94
bleeding sites
  Change from Baseline at Week 3: number analyzed (Participants) | 90
  Change from Baseline at Week 3 | -2.4 (1.02)
  Change from Baseline at Week 6: number analyzed (Participants) | 92
  Change from Baseline at Week 6 | -2.4 (1.26)
Statistical Analysis 1: Comparison: Test Product (Corsodyl Original Toothpaste); Change from Baseline at Week 3 (Test for non-zero within group change from Baseline); Test type: Superiority; p = 0.0181, MMRM
Statistical Analysis 2: Comparison: Test Product (Corsodyl Original Toothpaste); Change from Baseline at Week 6 (Test for non-zero within group change from Baseline); Test type: Superiority; p = 0.0541, MMRM

4. Secondary Outcome: Adjusted Mean Change From Baseline in Number of Bleeding Sites at Week 3 and Week 6 (Test Product vs. Reference Product)
Description: as for outcome 3
Time Frame: Baseline, Week 3, and Week 6
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Least Squares Mean (Standard Error); unit: bleeding sites
Arm/Group | Test Product (Corsodyl Original Toothpaste) | Reference Product (Colgate Cavity Protection Toothpaste)
Number analyzed (Participants) | 94 | 96
bleeding sites
  Change from Baseline at Week 3: number analyzed (Participants) | 90 | 91
  Change from Baseline at Week 3 | -2.4 (1.02) | 1.4 (1.02)
  Change from Baseline at Week 6: number analyzed (Participants) | 92 | 92
  Change from Baseline at Week 6 | -2.4 (1.26) | 2.9 (1.25)
Statistical Analysis 1: Comparison: Test Product (Corsodyl Original Toothpaste) vs Reference Product (Colgate Cavity Protection Toothpaste); Change from Baseline at Week 3; Test type: Superiority; p = 0.0091, MMRM; Adjusted Mean Difference = -3.8, 95% CI 2-sided [-6.7 to -1.0], Standard Error of Mean 1.44 — Adjusted mean difference was calculated as test product minus reference product
Statistical Analysis 2: Comparison: Test Product (Corsodyl Original Toothpaste) vs Reference Product (Colgate Cavity Protection Toothpaste); Change from Baseline at Week 6; Test type: Superiority; p = 0.0031, MMRM; Adjusted Mean Difference = -5.3, 95% CI 2-sided [-8.8 to -1.8], Standard Error of Mean 1.78 — Adjusted mean difference was calculated as test product minus reference product

5. Secondary Outcome: Adjusted Mean Change From Baseline in Mean BI at Weeks 3, 6 and 12
Description: The BI was assessed for all evaluable surfaces (having two-thirds of the natural tooth surface gradable for the assessment) of the facial and lingual/palatal gingiva, 6 sites per tooth (mesiobuccal, buccal, and distobuccal; mesiolingual/palatal, lingual/palatal, and distolingual/palatal). Evaluable tooth sites were probed, and gingival bleeding was assessed for approximately 30 seconds after probing and scored on a 3-point scale ranging from 0 to 2, where 0=No bleeding after 30 seconds; 1=Bleeding observed within 30 seconds of probing; 2=Bleeding observed immediately on probing. Mean BI was calculated by taking the average over all tooth sites assessed for a participant. Lower score indicated better outcome. Change from Baseline was calculated by subtracting the Baseline value from the value at each indicated timepoint. Baseline was defined as Day 0. A negative change from Baseline indicated improvement in gingival bleeding.
Time Frame: Baseline, Weeks 3, 6 and 12
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Product (Corsodyl Original Toothpaste)
Number analyzed (Participants) | 94
score on a scale
  Change from Baseline at Week 3: number analyzed (Participants) | 90
  Change from Baseline at Week 3 | -0.04 (0.008)
  Change from Baseline at Week 6: number analyzed (Participants) | 92
  Change from Baseline at Week 6 | -0.04 (0.009)
  Change from Baseline at Week 12: number analyzed (Participants) | 92
  Change from Baseline at Week 12 | -0.06 (0.011)
Statistical Analysis 1: Comparison: Test Product (Corsodyl Original Toothpaste); Change from Baseline at Week 3 (Test for non-zero within group change from Baseline); Test type: Superiority; p < 0.0001, MMRM
Statistical Analysis 2: Comparison: Test Product (Corsodyl Original Toothpaste); Change from Baseline at Week 6 (Test for non-zero within group change from Baseline); Test type: Superiority; p < 0.0001, MMRM
Statistical Analysis 3: Comparison: Test Product (Corsodyl Original Toothpaste); Change from Baseline at Week 12 (Test for non-zero within group change from Baseline); Test type: Superiority; p < 0.0001, MMRM

6. Secondary Outcome: Adjusted Mean Change From Baseline in Mean BI at Weeks 3, 6 and 12 (Test Product vs. Reference Product)
Description: as for outcome 5
Time Frame: Baseline, Weeks 3, 6 and 12
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Product (Corsodyl Original Toothpaste) | Reference Product (Colgate Cavity Protection Toothpaste)
Number analyzed (Participants) | 94 | 96
score on a scale
  Change from Baseline at Week 3: number analyzed (Participants) | 90 | 91
  Change from Baseline at Week 3 | -0.04 (0.008) | -0.01 (0.008)
  Change from Baseline at Week 6: number analyzed (Participants) | 92 | 92
  Change from Baseline at Week 6 | -0.04 (0.009) | -0.00 (0.009)
  Change from Baseline at Week 12: number analyzed (Participants) | 92 | 96
  Change from Baseline at Week 12 | -0.06 (0.011) | -0.01 (0.011)
Statistical Analysis 1: Comparison: Test Product (Corsodyl Original Toothpaste) vs Reference Product (Colgate Cavity Protection Toothpaste); Change from Baseline at Week 3; Test type: Superiority; p = 0.0051, MMRM; Adjusted Mean Difference = -0.03, 95% CI 2-sided [-0.05 to -0.01], Standard Error of Mean 0.011 — Adjusted mean difference was calculated as test product minus reference product
Statistical Analysis 2: Comparison: Test Product (Corsodyl Original Toothpaste) vs Reference Product (Colgate Cavity Protection Toothpaste); Change from Baseline at Week 6; Test type: Superiority; p = 0.0034, MMRM; Adjusted Mean Difference = -0.04, 95% CI 2-sided [-0.07 to -0.01], Standard Error of Mean 0.013 — Adjusted mean difference was calculated as test product minus reference product
Statistical Analysis 3: Comparison: Test Product (Corsodyl Original Toothpaste) vs Reference Product (Colgate Cavity Protection Toothpaste); Change from Baseline at Week 12; Test type: Superiority; p = 0.0022, MMRM; Adjusted Mean Difference = -0.05, 95% CI 2-sided [-0.08 to -0.02], Standard Error of Mean 0.015 — Adjusted mean difference was calculated as test product minus reference product

7. Secondary Outcome: Adjusted Mean Change From Baseline in Mean Mean Modified Gingival Index (MGI) at Weeks 3, 6 and 12
Description: MGI assessment is a non-invasive evaluation which focuses on visual symptoms of gingivitis (example, redness, texture, edema). MGI was assessed for all evaluable surfaces of facial and lingual/palatal gingiva,4 sites per tooth and scored on a 5-point scale ranging from 0 to 4, where 0=Absence of inflammation;1=Mild inflammation;slight change in color,little change in color;little change in texture of any portion of marginal or papillary gingival unit;2=Mild inflammation; criteria as 1 but involving the entire marginal or papillary gingival unit;3=Moderate inflammation;glazing, redness, edema, and/or hypertrophy of marginal or papillary gingival unit;4= Severe inflammation;marked redness, edema and/or hypertrophy of marginal or papillary gingival unit,spontaneous bleeding, congestion, or ulceration. Lower score indicated better outcome. Change from Baseline=Value at each indicated timepoint minus Baseline [Day 0] value. A negative change from Baseline indicated improvement in symptoms.
Time Frame: Baseline, Weeks 3, 6 and 12
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Product (Corsodyl Original Toothpaste)
Number analyzed (Participants) | 94
score on a scale
  Change from Baseline at Week 3: number analyzed (Participants) | 90
  Change from Baseline at Week 3 | -0.12 (0.014)
  Change from Baseline at Week 6: number analyzed (Participants) | 92
  Change from Baseline at Week 6 | -0.19 (0.019)
  Change from Baseline at Week 12: number analyzed (Participants) | 92
  Change from Baseline at Week 12 | -0.24 (0.021)
Statistical Analysis 1: Comparison: Test Product (Corsodyl Original Toothpaste); Change from Baseline at Week 3 (Test for non-zero within group change from Baseline); Test type: Superiority; p < 0.0001, MMRM
Statistical Analysis 2: Comparison: Test Product (Corsodyl Original Toothpaste); Change from Baseline at Week 6 (Test for non-zero within group change from Baseline); Test type: Superiority; p < 0.0001, MMRM
Statistical Analysis 3: Comparison: Test Product (Corsodyl Original Toothpaste); Change from Baseline at Week 12 (Test for non-zero within group change from Baseline); Test type: Superiority; p < 0.0001, MMRM

8. Secondary Outcome: Adjusted Mean Change From Baseline in Mean MGI at Weeks 3, 6 and 12 (Test Product vs. Reference Product)
Description: as for outcome 7
Time Frame: Baseline, Weeks 3, 6 and 12
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Product (Corsodyl Original Toothpaste) | Reference Product (Colgate Cavity Protection Toothpaste)
Number analyzed (Participants) | 94 | 96
score on a scale
  Change from Baseline at Week 3: number analyzed (Participants) | 90 | 91
  Change from Baseline at Week 3 | -0.12 (0.014) | -0.04 (0.014)
  Change from Baseline at Week 6: number analyzed (Participants) | 92 | 92
  Change from Baseline at Week 6 | -0.19 (0.019) | -0.06 (0.019)
  Change from Baseline at Week 12: number analyzed (Participants) | 92 | 96
  Change from Baseline at Week 12 | -0.24 (0.021) | -0.10 (0.021)
Statistical Analysis 1: Comparison: Test Product (Corsodyl Original Toothpaste) vs Reference Product (Colgate Cavity Protection Toothpaste); Change from Baseline at Week 3; Test type: Superiority; p < 0.0001, MMRM; Adjusted Mean Difference = -0.08, 95% CI 2-sided [-0.12 to -0.04], Standard Error of Mean 0.020 — Adjusted mean difference was calculated as test product minus reference product
Statistical Analysis 2: Comparison: Test Product (Corsodyl Original Toothpaste) vs Reference Product (Colgate Cavity Protection Toothpaste); Change from Baseline at Week 6; Test type: Superiority; p < 0.0001, MMRM; Adjusted Mean Difference = -0.12, 95% CI 2-sided [-0.18 to -0.07], Standard Error of Mean 0.027 — Adjusted mean difference was calculated as test product minus reference product
Statistical Analysis 3: Comparison: Test Product (Corsodyl Original Toothpaste) vs Reference Product (Colgate Cavity Protection Toothpaste); Change from Baseline at Week 12; Test type: Superiority; p < 0.0001, MMRM; Adjusted Mean Difference = -0.14, 95% CI 2-sided [-0.20 to -0.08], Standard Error of Mean 0.030 — Adjusted mean difference was calculated as test product minus reference product

9. Secondary Outcome: Adjusted Mean Change From Baseline in Mean Overall TPI (Turesky Plaque Index) at Weeks 3, 6 and 12
Description: TPI was used to assess plaque on the facial and lingual surfaces of each scorable tooth (7-7 in each arch). 3 scores were recorded facially(distal, body, mesial sites), and 3 scores were recorded lingually(distal, body, mesial sites). Plaque was first disclosed using a dye solution and scored on a 6-point scale ranging from 0 to 5, where 0=No plaque; 1=Separate flecks of plaque at the cervical margin; 2=Thin continuous band of plaque (up to 1 millimeter[mm]) at the cervical margin; 3=Band of plaque wider than 1 mm but covering less than (<)1/3 of the tooth surface; 4=Plaque covering greater than or equal to (>=)1/3 but <2/3 of the tooth surface; 5=Plaque covering >=2/3 of the tooth surface. Mean overall TPI score=Average of TPI values over all tooth sites assessed for a participant. Lower score=better outcome. Change from Baseline=Value at each indicated timepoint minus Baseline value. Baseline=Day 0. A negative change from Baseline indicated improvement (less plaque accumulation).
Time Frame: Baseline, Weeks 3, 6 and 12
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Product (Corsodyl Original Toothpaste)
Number analyzed (Participants) | 94
score on a scale
  Change from Baseline at Week 3: number analyzed (Participants) | 90
  Change from Baseline at Week 3 | -0.32 (0.033)
  Change from Baseline at Week 6: number analyzed (Participants) | 92
  Change from Baseline at Week 6 | -0.31 (0.043)
  Change from Baseline at Week 12: number analyzed (Participants) | 92
  Change from Baseline at Week 12 | -0.41 (0.047)
Statistical Analysis 1: Comparison: Test Product (Corsodyl Original Toothpaste); Change from Baseline at Week 3 (Test for non-zero within group change from Baseline); Test type: Superiority; p < 0.0001, MMRM
Statistical Analysis 2: Comparison: Test Product (Corsodyl Original Toothpaste); Change from Baseline at Week 6 (Test for non-zero within group change from Baseline); Test type: Superiority; p < 0.0001, MMRM
Statistical Analysis 3: Comparison: Test Product (Corsodyl Original Toothpaste); Change from Baseline at Week 12 (Test for non-zero within group change from Baseline); Test type: Superiority; p < 0.0001, MMRM

10. Secondary Outcome: Adjusted Mean Change From Baseline in Mean Overall TPI at Weeks 3, 6 and 12 (Test Product vs. Reference Product)
Description: TPI was used to assess plaque on the facial and lingual surfaces of each scorable tooth (7-7 in each arch). 3 scores were recorded facially (distal, body, mesial sites), and 3 scores were recorded lingually (distal, body, mesial sites). Plaque was first disclosed using a dye solution and scored on a 6-point scale ranging from 0 to 5, where 0=No plaque; 1=Separate flecks of plaque at the cervical margin; 2=Thin continuous band of plaque (up to 1 mm) at the cervical margin; 3=Band of plaque wider than 1 mm but covering <1/3 of the tooth surface; 4=Plaque covering >=1/3 but <2/3 of the tooth surface; 5=Plaque covering >=2/3 of the tooth surface. Mean overall TPI score=Average of TPI values over all tooth sites assessed for a participant. Lower score=better outcome. Change from Baseline=Value at each indicated timepoint minus Baseline value. Baseline=Day 0. A negative change from Baseline indicated improvement (less plaque accumulation).
Time Frame: Baseline, Weeks 3, 6 and 12
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Product (Corsodyl Original Toothpaste) | Reference Product (Colgate Cavity Protection Toothpaste)
Number analyzed (Participants) | 94 | 96
score on a scale
  Change from Baseline at Week 3: number analyzed (Participants) | 90 | 91
  Change from Baseline at Week 3 | -0.32 (0.033) | -0.17 (0.033)
  Change from Baseline at Week 6: number analyzed (Participants) | 92 | 92
  Change from Baseline at Week 6 | -0.31 (0.043) | -0.14 (0.043)
  Change from Baseline at Week 12: number analyzed (Participants) | 92 | 96
  Change from Baseline at Week 12 | -0.41 (0.047) | -0.12 (0.046)
Statistical Analysis 1: Comparison: Test Product (Corsodyl Original Toothpaste) vs Reference Product (Colgate Cavity Protection Toothpaste); Change from Baseline at Week 3; Test type: Superiority; p = 0.0012, MMRM; Adjusted Mean Difference = -0.15, 95% CI 2-sided [-0.25 to -0.06], Standard Error of Mean 0.047 — Adjusted mean difference was calculated as test product minus reference product
Statistical Analysis 2: Comparison: Test Product (Corsodyl Original Toothpaste) vs Reference Product (Colgate Cavity Protection Toothpaste); Change from Baseline at Week 6; Test type: Superiority; p = 0.0058, MMRM; Adjusted Mean Difference = -0.17, 95% CI 2-sided [-0.29 to -0.05], Standard Error of Mean 0.061 — Adjusted mean difference was calculated as test product minus reference product
Statistical Analysis 3: Comparison: Test Product (Corsodyl Original Toothpaste) vs Reference Product (Colgate Cavity Protection Toothpaste); Change from Baseline at Week 12; Test type: Superiority; p < 0.0001, MMRM; Adjusted Mean Difference = -0.29, 95% CI 2-sided [-0.42 to -0.16], Standard Error of Mean 0.066 — Adjusted mean difference was calculated as test product minus reference product

11. Secondary Outcome: Adjusted Mean Change From Baseline in Mean Interproximal TPI at Weeks 3, 6 and 12
Description: TPI was used to assess plaque on the facial and lingual surfaces of each scorable tooth (7-7 in each arch). 3 scores were recorded facially (distal, mesial sites), and 3 scores were recorded lingually (distal, mesial sites). Plaque was first disclosed using a dye solution and scored on a 6-point scale ranging from 0 to 5, where 0=No plaque; 1=Separate flecks of plaque at the cervical margin; 2=Thin continuous band of plaque (up to 1 mm) at the cervical margin; 3=Band of plaque wider than 1 mm but covering <1/3 of the tooth surface; 4=Plaque covering >=1/3 but <2/3 of the tooth surface; 5=Plaque covering >=2/3 of the tooth surface. Mean interproximal TPI score=Average of TPI values over distal and mesial tooth sites assessed for a participant. Lower score indicated better outcome. Change from Baseline=Value at each indicated timepoint minus Baseline value. Baseline=Day 0. A negative change from Baseline indicated improvement (less plaque accumulation).
Time Frame: Baseline, Weeks 3, 6 and 12
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Product (Corsodyl Original Toothpaste)
Number analyzed (Participants) | 94
score on a scale
  Change from Baseline at Week 3: number analyzed (Participants) | 90
  Change from Baseline at Week 3 | -0.35 (0.036)
  Change from Baseline at Week 6: number analyzed (Participants) | 92
  Change from Baseline at Week 6 | -0.34 (0.047)
  Change from Baseline at Week 12: number analyzed (Participants) | 92
  Change from Baseline at Week 12 | -0.42 (0.052)
Statistical Analysis 1: Comparison: Test Product (Corsodyl Original Toothpaste); Change from Baseline at Week 3 (Test for non-zero within group change from Baseline); Test type: Superiority; p < 0.0001, MMRM
Statistical Analysis 2: Comparison: Test Product (Corsodyl Original Toothpaste); Change from Baseline at Week 6 (Test for non-zero within group change from Baseline); Test type: Superiority; p < 0.0001, MMRM
Statistical Analysis 3: Comparison: Test Product (Corsodyl Original Toothpaste); Change from Baseline at Week 12 (Test for non-zero within group change from Baseline); Test type: Superiority; p < 0.0001, MMRM

12. Secondary Outcome: Adjusted Mean Change From Baseline in Mean Interproximal TPI at Weeks 3, 6 and 12 (Test Product vs. Reference Product)
Description: as for outcome 11
Time Frame: Baseline, Weeks 3, 6 and 12
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Product (Corsodyl Original Toothpaste) | Reference Product (Colgate Cavity Protection Toothpaste)
Number analyzed (Participants) | 94 | 96
score on a scale
  Change from Baseline at Week 3: number analyzed (Participants) | 90 | 91
  Change from Baseline at Week 3 | -0.35 (0.036) | -0.19 (0.036)
  Change from Baseline at Week 6: number analyzed (Participants) | 92 | 92
  Change from Baseline at Week 6 | -0.34 (0.047) | -0.17 (0.047)
  Change from Baseline at Week 12: number analyzed (Participants) | 92 | 96
  Change from Baseline at Week 12 | -0.42 (0.052) | -0.12 (0.052)
Statistical Analysis 1: Comparison: Test Product (Corsodyl Original Toothpaste) vs Reference Product (Colgate Cavity Protection Toothpaste); Change from Baseline at Week 3; Test type: Superiority; p = 0.0022, MMRM; Adjusted Mean Difference = -0.16, 95% CI 2-sided [-0.26 to -0.06], Standard Error of Mean 0.051 — Adjusted mean difference was calculated as test product minus reference product
Statistical Analysis 2: Comparison: Test Product (Corsodyl Original Toothpaste) vs Reference Product (Colgate Cavity Protection Toothpaste); Change from Baseline at Week 6; Test type: Superiority; p = 0.0099, MMRM; Adjusted Mean Difference = -0.17, 95% CI 2-sided [-0.30 to -0.04], Standard Error of Mean 0.066 — Adjusted mean difference was calculated as test product minus reference product
Statistical Analysis 3: Comparison: Test Product (Corsodyl Original Toothpaste) vs Reference Product (Colgate Cavity Protection Toothpaste); Change from Baseline at Week 12; Test type: Superiority; p < 0.0001, MMRM; Adjusted Mean Difference = -0.30, 95% CI 2-sided [-0.45 to -0.16], Standard Error of Mean 0.073 — Adjusted mean difference was calculated as test product minus reference product

ADVERSE EVENTS:
Time Frame: From signing of informed consent form until 5 days after last administration of study product or last study procedure (up to approximately 111 days)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of one of the study products including any washout or lead-in product (or medical device), whether or not considered related to the study product, including any washout or lead-in product (or medical device). A Serious Adverse Event (SAE) was a particular category of an AE where the adverse outcome is serious.
Arm/Group | Test Product (Corsodyl Original Toothpaste) | Reference Product (Colgate Cavity Protection Toothpaste)
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/96
Other Adverse Events (participants affected / at risk) | 2/94 | 4/96
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Product (Corsodyl Original Toothpaste) (N=94) | Reference Product (Colgate Cavity Protection Toothpaste) (N=96)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 | 1
TOOTHACHE (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 1
GINGIVAL INJURY (Injury, poisoning and procedural complications) | 2 | 0
MIGRAINE (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT05654662/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/62/NCT05654662/SAP_001.pdf